CLINICAL TRIAL: NCT00081770
Title: Comparison of PEG-Intron 1.5µg/kg/wk Plus REBETOL vs PEG-Intron 1µg/kg/wk Plus REBETOL vs PEGASYS 180µg/wk Plus COPEGUS in Previously Untreated Adult Subjects With Chronic Hepatitis C Infected With Genotype 1
Brief Title: Peginterferon Dose Evaluations for Previously Untreated Subjects With Chronic Hepatitis C Infected With Genotype 1 (Study P03471)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03471; 2552898
Record Dates: First submitted 2004-04-20; First posted 2004-04-22 (Estimated); Results first posted 2009-10-30 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PegIntron 1.5 ug/kg/wk plus REBETOL (Experimental): PegIntron (peginterferon alfa-2b; SCH 54031) 1.5 ug/kg/week in combination with weight-based REBETOL (ribavirin; SCH 18908) 800-1400 mg/day administered for 48 weeks with 24-week post-treatment follow-up
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: REBETOL (ribavirin; SCH 18908)
- PegIntron 1.0 ug/kg/wk plus REBETOL (Experimental): PegIntron (peginterferon alfa-2b; SCH 54031) 1.0 ug/kg/week in combination with weight-based REBETOL (ribavirin; SCH 18908) 800-1400 mg/day administered for 48 weeks with 24-week post-treatment follow-up
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: REBETOL (ribavirin; SCH 18908)
- PEGASYS 180 ug/wk Plus COPEGUS (Active Comparator): PEGASYS (peginterferon alfa-2a) 180 ug/week plus COPEGUS (ribavirin) 1000-1200 mg/day administered for 48 weeks with 24-week post-treatment follow-up
  Interventions: Biological: PEGASYS (peginterferon alfa-2a); Drug: COPEGUS (ribavirin)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — 1.5 ug/kg/week subcutaneously (SC) for 48 weeks
  Other Names: PegIntron
  Arms: PegIntron 1.5 ug/kg/wk plus REBETOL
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — 1.0 ug/kg/week SC for 48 weeks
  Other Names: PegIntron
  Arms: PegIntron 1.0 ug/kg/wk plus REBETOL
Drug: REBETOL (ribavirin; SCH 18908) — weight based dose 800-1400 mg/day orally (PO) for 48 weeks
  Other Names: REBETOL [the Schering-Plough brand name for ribavirin]
  Arms: PegIntron 1.0 ug/kg/wk plus REBETOL; PegIntron 1.5 ug/kg/wk plus REBETOL
Biological: PEGASYS (peginterferon alfa-2a) — 180 ug/week SC administered for 48 weeks
  Other Names: PEGASYS
  Arms: PEGASYS 180 ug/wk Plus COPEGUS
Drug: COPEGUS (ribavirin) — 1000-1200 mg/day PO for 48 weeks
  Other Names: COPEGUS [the Hoffman-La Roche brand name for ribavirin]
  Arms: PEGASYS 180 ug/wk Plus COPEGUS

SUMMARY:
The objective is to compare the safety and efficacy of the following three treatment regimens in previously untreated adult subjects with chronic hepatitis C infected with Genotype 1: (1) PegIntron 1.5 µg/kg/wk in combination with weight based REBETOL (800-1400 mg/day); (2) PegIntron 1µg/kg/wk in combination with weight based REBETOL (800-1400 mg/day); and (3) PEGASYS 180 µg/wk plus COPEGUS 1000-1200 mg/day.

DETAILED DESCRIPTION:
PegIntron Dose will be administered once weekly subcutaneously on the same day of the week:

Screening 2 Weight 40-50 kg Volume to Inject (mL) 0.22; Screening 2 Weight 51-60 kg Volume to Inject (mL) 0.28; Screening 2 Weight 61-75 kg Volume to Inject (mL) 0.33; Screening 2 Weight 76-85 kg Volume to Inject (mL) 0.41; Screening 2 Weight 86-104 kg Volume to Inject (mL) 0.48; Screening 2 Weight 105-125 kg Volume to Inject (mL) 0.58 from two vials

REBETOL Dosage (for Use With PegIntron):

Screening 2 Weight 40-65 kg Daily Dose 800 mg; Screening 2 Weight >65-85 kg Daily Dose 1000 mg; Screening 2 Weight >85-105 kg Daily Dose 1200 mg; Screening 2 Weight >105-125 kg Daily Dose 1400 mg

The PEGASYS dose of 1 mL (180 µg) will be administered once weekly subcutaneously on the same day of the week

COPEGUS Dosage (for Use With PEGASYS):

Screening 2 Weight <75 kg Daily Dose 1000 mg; Screening 2 Weight > or = 75 kg Daily Dose 1200mg

NOTE: Double Blind for PegIntron; Open Label for REBETOL, PEGASYS and COPEGUS

NOTE: REBETOL is the Schering-Plough brand name for ribavirin. COPEGUS is the Hoffman-La Roche brand name for ribavirin.

ELIGIBILITY:
INCLUSION CRITERIA:

* Previously untreated adults with chronic hepatitis C (hepatitis C virus ribonucleic acid [HCV RNA] quantitative polymerase chain reaction [qPCR] plasma positive)
* Individuals with HCV genotype 1 (mixed 1a/1b is acceptable)
* Compensated liver disease
* Pretreatment liver biopsy slides available
* Adults aged 18-70
* Individuals weighing 88-275 pounds (40-125 kg)
* Free from substance abuse for past 2 years
* Those suffering from diabetes and/or hypertension must have normal eye exams and retinal photographs (these will be done as part of the study before hepatitis C treatment is given)
* Patients and partners of patients willing to use adequate contraception during the course of the study
* Hematology laboratory results of:

  * Hemoglobin (HGB) ≥ 12 g/dL for females or ≥ 13g/dL for males
  * White Blood Cell Count (WBC) ≥ 3,000/mm^3
  * Neutrophils ≥ 1,500/mm^3
  * Platelets ≥ 80,000/mm^3
* Chemistry laboratory results of:

  * Normal Thyroid Stimulating Hormone (TSH), albumin, creatinine, and direct bilirubin
  * Antinuclear antibody (ANA) ≤ 1:320
  * Fasting Glucose 70-140 mg/dL Note: If glucose levels are between 116-140 mg/dL or an individual has diabetes, glycosylated hemoglobin [HbA1C] must be ≤ 8.5%

EXCLUSION CRITERIA:

* Previous hepatitis C treatment
* Pregnant women or partners of pregnant women
* Patients or partners of patients who intend to become pregnant any time during the 48 weeks
* Women who are breastfeeding
* Individuals with liver disease not caused by hepatitis C
* Individuals infected with the hepatitis B virus and/or human immunodeficiency virus (HIV)
* Patients with a history of liver cancer (hepatocellular carcinoma)
* Known blood disorders such as hemoglobinopathy, coagulopathy, or glucose-6-phosphate dehydrogenase [G6PD] deficiency
* Body organ transplant
* Any known or suspected cancer within the past 5 years
* Individuals who currently use epoetin [EPO], granulocyte colony stimulating factor [G-CSF] and/or granulocyte monocyte colony stimulating factor [GM-CSF]
* Those having a history of or active clinical gout
* Individuals who have chronic pulmonary disease
* Individuals who have a medical condition that would likely require systemic steroids
* Those with a history of central nervous system (CNS trauma) or seizure disorders
* Current or previous use of lithium or antipsychotic drugs
* Individuals who currently have or show signs of moderate to severe depression or history of significant psychiatric disorders
* Patients with clinically significant electrocardiogram (ECG) abnormalities
* Individuals with serious heart problems such as those who have had a heart attack, uncontrolled high blood pressure, or other heart problems
* Patients that weigh > 231-275 pounds (105-125 kg) AND have a body mass index (BMI) > 30 AND have 3 or more of the risk factors below: (a) Strong family history of coronary heart disease (CHD) which includes 2 or more first-degree relatives with CHD or family history of early CHD at age < 55 for male relatives or < 65 for female relatives (b) Individuals with abnormal total cholesterol and/or sub fractions (uncontrolled hypercholesterolemia) (c) Diabetes (d) Hypertension (e) Smoking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4469 (Actual)
Dates: Start 2004-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] McHutchison JG, Lawitz EJ, Shiffman ML, Muir AJ, Galler GW, McCone J, Nyberg LM, Lee WM, Ghalib RH, Schiff ER, Galati JS, Bacon BR, Davis MN, Mukhopadhyay P, Koury K, Noviello S, Pedicone LD, Brass CA, Albrecht JK, Sulkowski MS; IDEAL Study Team. Peginterferon alfa-2b or alfa-2a with ribavirin for treatment of hepatitis C infection. N Engl J Med. 2009 Aug 6;361(6):580-93. doi: 10.1056/NEJMoa0808010. Epub 2009 Jul 22. PMID 19625712
- [Derived] Melia MT, Muir AJ, McCone J, Shiffman ML, King JW, Herrine SK, Galler GW, Bloomer JR, Nunes FA, Brown KA, Mullen KD, Ravendhran N, Ghalib RH, Boparai N, Jiang R, Noviello S, Brass CA, Albrecht JK, McHutchison JG, Sulkowski MS; IDEAL Study Team. Racial differences in hepatitis C treatment eligibility. Hepatology. 2011 Jul;54(1):70-8. doi: 10.1002/hep.24358. PMID 21488082

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled 4469 subjects; Randomized 3083; Treated 3070
Period: Overall Study
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS
Started | 1019 | 1016 | 1035
Completed | 517 (Patients who discontinued treatment but continued in study are considered Not Completed) | 470 (Patients who discontinued treatment but continued in study are considered Not Completed) | 579 (Patients who discontinued treatment but continued in study are considered Not Completed)
Not Completed | 502 | 546 | 456
Not completed — Adverse Event | 130 | 98 | 136
Not completed — Lack of Efficacy | 262 | 357 | 211
Not completed — Lost to Follow-up | 45 | 34 | 45
Not completed — Protocol Violation | 15 | 10 | 10
Not completed — Withdrawal by Subject | 45 | 40 | 42
Not completed — Did not meet protocol eligibility | 2 | 0 | 3
Not completed — Administrative | 1 | 0 | 1
Not completed — Other | 2 | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS | Total
Number analyzed (Participants) | 1019 | 1016 | 1035 | 3070
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (7.8) | 47.5 (8.1) | 47.6 (8.2) | 47.5 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 406 | 409 | 422 | 1237
  Male | 613 | 607 | 613 | 1833

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR) Rate
Description: SVR rate is the percentage of participants with undetectable hepatitis C virus ribonucleic acid (HCV-RNA) at the end of the 24-week post-treatment follow-up.
Time Frame: Assessed at the end of a 24-week post-treatment follow-up
Population: Intent-to-Treat [ITT] Population defined as subjects who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS
Number analyzed (Participants) | 1019 | 1016 | 1035
Percentage of participants | 39.8 | 38.0 | 40.9
Statistical Analysis 1: Comparison: PegIntron 1.5 ug/kg/wk Plus REBETOL vs PEGASYS 180 ug/wk Plus COPEGUS; Test type: Superiority or Other; p = 0.567, Regression, Logistic — Holm's method for multiplicity adjustment was to be used to control the overall Type I error rate at α = 0.05. However, since there was no significant difference in the overall SVR rates between the three groups, no Type-1 error adjustment was made; The p-value is based on the logistic regression model that includes treatment and baseline stratification factors (viral load and race); Odds Ratio (OR) = 0.95, 95% CI [0.79 to 1.14] — The odds ratio is based on the logistic regression model that includes treatment and baseline stratification factors: viral load (≤600,000 IU/mL vs >600,000 IU/mL) and race (Black vs non-Black)
Statistical Analysis 2: Comparison: PegIntron 1.5 ug/kg/wk Plus REBETOL vs PegIntron 1.0 ug/kg/wk Plus REBETOL; Test type: Superiority or Other; p = 0.195, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.08, 95% CI [0.90 to 1.30] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean Change From Baseline in the Log Viral Load at Treatment Week 4
Description: The difference between viral load levels in the blood at the start of the study and Treatment Week 4, expressed in terms of a logarithmic scale with base 10, and averaged for all the participants in each treatment group.
Time Frame: Assessed at Baseline and Treatment Week 4
Population: ITT Population defined as subjects who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS
Number analyzed (Participants) | 1019 | 1016 | 1035
Log10 IU/mL | -2.32 (1.50) | -2.02 (1.42) | -2.45 (1.52)

3. Secondary Outcome: Virologic Response Rate at Treatment Week 12
Description: Percentage of participants with undetectable hepatitis C RNA (HCV-RNA) at Treatment Week 12
Time Frame: Assessed at Treatment Week 12
Population: ITT Population defined as subjects who received at least one dose of study medication
Measure: Number; unit: Percentage of participants
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS
Number analyzed (Participants) | 1019 | 1016 | 1035
Percentage of participants | 39.9 | 36.0 | 45.0
Statistical Analysis 1: Comparison: PegIntron 1.5 ug/kg/wk Plus REBETOL; Test type: Superiority or Other; Percentage of participants = 39.9, 95% CI [36.9 to 42.9] — Percentage of participants with undetectable HCV-RNA at Treatment Week 12
Statistical Analysis 2: Comparison: PegIntron 1.0 ug/kg/wk Plus REBETOL; Test type: Superiority or Other; Percentage of participants = 36.0, 95% CI [33.1 to 39.0] — Percentage of participants with undetectable HCV-RNA at Treatment Week 12
Statistical Analysis 3: Comparison: PEGASYS 180 ug/wk Plus COPEGUS; Test type: Superiority or Other; Percentage of participants = 45.0, 95% CI [42.0 to 48.1] — Percentage of participants with undetectable HCV-RNA at Treatment Week 12

4. Secondary Outcome: Mean Change From Baseline in the Log Viral Load at Treatment Week 2
Description: The difference between viral load levels in the blood at the start of the study and Treatment Week 2, expressed in terms of a logarithmic scale with base 10, and averaged for all the participants in each treatment group.
Time Frame: Assessed at Baseline and Treatment Week 2
Population: ITT Population defined as subjects who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: Log10 IU/mL
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS
Number analyzed (Participants) | 1019 | 1016 | 1035
Log10 IU/mL | -1.55 (1.20) | -1.30 (1.12) | -1.60 (1.24)

ADVERSE EVENTS:
Arm/Group | PegIntron 1.5 ug/kg/wk Plus REBETOL | PegIntron 1.0 ug/kg/wk Plus REBETOL | PEGASYS 180 ug/wk Plus COPEGUS
Serious Adverse Events (participants affected / at risk) | 88/1019 | 94/1016 | 121/1035
Other Adverse Events (participants affected / at risk) | 996/1019 | 1000/1016 | 1018/1035
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron 1.5 ug/kg/wk Plus REBETOL (N=1019) | PegIntron 1.0 ug/kg/wk Plus REBETOL (N=1016) | PEGASYS 180 ug/wk Plus COPEGUS (N=1035)
ANAEMIA (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 1 (1)
APLASTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
LYMPHADENITIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CORONARY ARTERY RESTENOSIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CYANOSIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2)
PALPITATIONS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
WOLFF-PARKINSON-WHITE SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
MACULOPATHY (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
PAPILLOEDEMA (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (3) | 4 (5) | 4 (4)
APPENDICITIS PERFORATED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
IRRITABLE BOWEL SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 5 (5)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATIC CYST (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATIC ENLARGEMENT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATIC MASS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
SALIVARY DUCT OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 3 (3) | 4 (4)
CHEST DISCOMFORT (General disorders) | 0 (0) | 2 (2) | 3 (3)
CHEST PAIN (General disorders) | 8 (8) | 8 (8) | 8 (8)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 (0) | 1 (1) | 0 (0)
FACE OEDEMA (General disorders) | 0 (0) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
HERNIA OBSTRUCTIVE (General disorders) | 0 (0) | 0 (0) | 1 (1)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 2 (2) | 1 (1)
PYREXIA (General disorders) | 2 (2) | 2 (2) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 3 (3) | 1 (1) | 1 (1)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 5 (5) | 3 (3) | 3 (3)
JAUNDICE (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
PORTAL HYPERTENSIVE GASTROPATHY (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
SARCOIDOSIS (Immune system disorders) | 2 (2) | 1 (1) | 3 (3)
ABDOMINAL WALL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ANOGENITAL WARTS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 2 (2) | 4 (4) | 4 (5)
BLASTOMYCOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BURSITIS INFECTIVE STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 2 (2) | 5 (5) | 6 (6)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
FOLLICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES OESOPHAGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
INFECTIVE TENOSYNOVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INJECTION SITE ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
KIDNEY INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
LOBAR PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
LUNG ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
PERITONEAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 2 (2) | 3 (3) | 6 (6)
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
SEPSIS SYNDROME (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
BACK INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
CONCUSSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
DRUG TOXICITY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HEAD INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
HUMAN BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (3) | 0 (0)
LUNG INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL BILE LEAK (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM ST SEGMENT DEPRESSION (Investigations) | 0 (0) | 0 (0) | 1 (1)
GRIP STRENGTH DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (1)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 3 (3)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
JOINT INSTABILITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
WEIGHT BEARING DIFFICULTY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
ACOUSTIC NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 2 (2)
HAEMANGIOMA OF LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
MALIGNANT NEOPLASM OF AMPULLA OF VATER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
AKATHISIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ANOXIC ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
COMA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CONVULSION (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
FACIAL PALSY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
PARAPLEGIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
PERONEAL NERVE PALSY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SPINAL CORD INFARCTION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
SYNCOPE (Nervous system disorders) | 4 (4) | 1 (1) | 3 (3)
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3) | 0 (0)
ACUTE PSYCHOSIS (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ANGER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
ANXIETY (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1)
COMPLETED SUICIDE (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0)
DEPENDENCE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 5 (9) | 3 (3) | 3 (3)
DISORIENTATION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
DRUG ABUSE (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
DRUG DEPENDENCE (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
HALLUCINATION, VISUAL (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
HOMICIDAL IDEATION (Psychiatric disorders) | 2 (3) | 2 (2) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
PARANOIA (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 13 (17) | 8 (8) | 5 (5)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
BLADDER DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CALCULUS URETERIC (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
RENAL PAIN (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
URINARY INCONTINENCE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
CERVICAL DYSPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
RECTOCELE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 2 (3)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 3 (3)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY SARCOIDOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
PHYSICAL ASSAULT (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
CYSTOPEXY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
HYSTERECTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 1 (1)
RECTOCELE REPAIR (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
SALPINGO-OOPHORECTOMY UNILATERAL (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
SPINAL FUSION SURGERY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegIntron 1.5 ug/kg/wk Plus REBETOL (N=1019) | PegIntron 1.0 ug/kg/wk Plus REBETOL (N=1016) | PEGASYS 180 ug/wk Plus COPEGUS (N=1035)
ANAEMIA (Blood and lymphatic system disorders) | 344 (555) | 291 (442) | 348 (556)
LEUKOPENIA (Blood and lymphatic system disorders) | 95 (153) | 69 (109) | 106 (206)
NEUTROPENIA (Blood and lymphatic system disorders) | 263 (466) | 188 (300) | 325 (670)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 29 (38) | 24 (45) | 64 (111)
HYPOTHYROIDISM (Endocrine disorders) | 56 (61) | 39 (42) | 48 (51)
VISION BLURRED (Eye disorders) | 46 (52) | 62 (69) | 74 (76)
ABDOMINAL PAIN (Gastrointestinal disorders) | 47 (59) | 53 (60) | 61 (70)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 51 (60) | 50 (55) | 54 (69)
CONSTIPATION (Gastrointestinal disorders) | 77 (85) | 83 (89) | 63 (68)
DIARRHOEA (Gastrointestinal disorders) | 170 (221) | 193 (230) | 173 (207)
DRY MOUTH (Gastrointestinal disorders) | 58 (60) | 53 (53) | 50 (52)
DYSPEPSIA (Gastrointestinal disorders) | 60 (62) | 62 (72) | 69 (78)
NAUSEA (Gastrointestinal disorders) | 433 (517) | 377 (462) | 375 (434)
VOMITING (Gastrointestinal disorders) | 150 (190) | 122 (149) | 119 (141)
ASTHENIA (General disorders) | 51 (57) | 44 (48) | 41 (43)
CHILLS (General disorders) | 397 (428) | 365 (421) | 243 (266)
FATIGUE (General disorders) | 672 (798) | 676 (802) | 656 (809)
INFLUENZA LIKE ILLNESS (General disorders) | 164 (203) | 154 (175) | 160 (182)
INJECTION SITE ERYTHEMA (General disorders) | 166 (172) | 178 (197) | 123 (125)
INJECTION SITE REACTION (General disorders) | 102 (118) | 112 (116) | 58 (62)
IRRITABILITY (General disorders) | 256 (317) | 262 (319) | 262 (314)
PAIN (General disorders) | 126 (156) | 138 (168) | 100 (124)
PYREXIA (General disorders) | 356 (417) | 331 (381) | 237 (264)
BRONCHITIS (Infections and infestations) | 34 (37) | 32 (39) | 60 (66)
SINUSITIS (Infections and infestations) | 59 (72) | 43 (53) | 72 (90)
WEIGHT DECREASED (Investigations) | 138 (164) | 105 (122) | 102 (116)
ANOREXIA (Metabolism and nutrition disorders) | 121 (131) | 96 (100) | 76 (81)
DECREASED APPETITE (Metabolism and nutrition disorders) | 184 (197) | 159 (167) | 142 (152)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 238 (296) | 237 (294) | 250 (307)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 105 (118) | 106 (125) | 120 (136)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 53 (64) | 51 (63) | 72 (88)
MYALGIA (Musculoskeletal and connective tissue disorders) | 274 (309) | 270 (305) | 233 (263)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 52 (55) | 56 (66) | 74 (105)
DISTURBANCE IN ATTENTION (Nervous system disorders) | 72 (81) | 53 (60) | 71 (81)
DIZZINESS (Nervous system disorders) | 172 (218) | 154 (194) | 145 (171)
DYSGEUSIA (Nervous system disorders) | 80 (88) | 73 (76) | 66 (70)
HEADACHE (Nervous system disorders) | 508 (646) | 486 (609) | 438 (559)
ANXIETY (Psychiatric disorders) | 114 (142) | 117 (143) | 112 (125)
DEPRESSION (Psychiatric disorders) | 259 (351) | 197 (263) | 215 (257)
INSOMNIA (Psychiatric disorders) | 401 (482) | 389 (460) | 428 (500)
COUGH (Respiratory, thoracic and mediastinal disorders) | 167 (202) | 183 (223) | 210 (256)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 176 (200) | 173 (201) | 172 (194)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 55 (58) | 55 (59) | 75 (81)
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 63 (69) | 67 (73) | 76 (86)
ALOPECIA (Skin and subcutaneous tissue disorders) | 233 (249) | 205 (211) | 176 (178)
DRY SKIN (Skin and subcutaneous tissue disorders) | 122 (134) | 117 (125) | 137 (162)
PRURITUS (Skin and subcutaneous tissue disorders) | 163 (194) | 138 (168) | 182 (222)
RASH (Skin and subcutaneous tissue disorders) | 225 (289) | 223 (280) | 290 (429)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less